CLINICAL TRIAL: NCT04248127
Title: The Influence of Honey-flavored Yogurt on Low-grade Inflammation and Gut Health in Middle to Older Aged Women.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1492622
Record Dates: First submitted 2019-11-04; First posted 2020-01-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Overweight
Keywords: Phenolic; Honey; Inflammation; Yogurt; Microbiome
MeSH Terms: conditions — Overweight; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized single-blind 2-arm crossover trial. Each arm will be 4 weeks in length, with a 4 week washout between arms.
Who Masked: Participant
Masking Description: The honey intervention or isocaloric amounts of sugar will be provided in yogurt. The study participant will not be told what sweetener they will be receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey sweetened yogurt (Experimental): 1 tbsp. of honey in 0.6 cup (150g) of plain yogurt. The participants will be asked to consume 2 morning servings of the yogurt for a total of 2 tbsp. of the assigned honey per day.
  Interventions: Other: Honey sweetened yogurt
- Sugar sweetened yogurt (Placebo Comparator): Sugar will be added to 0.6 cup (150g) of plain yogurt in an isocaloric amount compared to the honey. The participants will be asked to consume 2 morning servings of the yogurt per day.
  Interventions: Other: Sugar sweetened yogurt

INTERVENTIONS:
Other: Honey sweetened yogurt — 2 tbsp. of daily honey intake in 1.2 cups of yogurt per day, split into two equal portions
  Arms: Honey sweetened yogurt
Other: Sugar sweetened yogurt — sugar added, in an isocaloric fashion to the honey, to 1.2 cups of yogurt per day, split into two equal portions
  Arms: Sugar sweetened yogurt

SUMMARY:
A randomized, double-blind, crossover dietary intervention trial will test the effects of 4 weeks of daily honey-flavored yogurt intake on markers of inflammation (Th17 cytokines) and oxidative stress (NOX2, UA, RSNO) and associative changes with microbial derived metabolites (SCFAs, BAs, ellagitannins), metabolism and the fecal microbiome. The above suite of selected markers will capture diet-induced systemic changes in inflammation and oxidative stress, while assessing associated microbial changes.

DETAILED DESCRIPTION:
Those qualified for enrollment will be randomized into a double-blind crossover study to consume 2 morning servings of a 0.6 cup (150g) of plain yogurt with : A) cane sugar added in an isocaloric level as the honey or, B) 1 tbsp of phenolic-rich honey for 4 weeks. A one-month washout between periods will be used. The participants will be instructed to consume one yogurt in replacement of or as part of breakfast, and as a late morning snack. They will also be instructed to not add any additional items to the yogurt. Therefore, each study participant will consume 2 tbsp. of honey a day for four weeks, which is a realistic amount typically consumed by honey users.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female: 45-65 years
* Women: lack of menses for at least two years.
* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures
* BMI 25.0 - 30.0 kg/m2

Exclusion Criteria:

* BMI ≥ 31 kg/m2
* Food allergies
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Use of concentrated food supplements/powders and extracts
* Fruit consumption > 2 cups/day
* Vegetable consumption >3 cups/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and stroke
* Abnormal Metabolic or CBC panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Currently taking prescription drugs or supplements.
* Supplement use other than a general formula of vitamins and minerals that meet the RDA
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* Cannabis use
* Screening LDL ≥ 190 mg/dl for those who have 0-1 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL]. (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp)
* Screening LDL ≥ 160 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL]. (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp);
* Screening LDL ≥ 130 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL], and a Framingham 10-year Risk Score 10-20% (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp).
* Current enrollee in a clinical research study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of CD4+ T Helper (TH)17 cytokines | 4 weeks
  Cytokines included in the panel are: Il-1b, IL-4, IL-6, IL-10, IL-17a, IL-21, IL-22, IL-23, IL-31, IL-33, IFN-gamma, TNF-alpha, IL-17f.

SECONDARY OUTCOMES:
Concentration of Secondary bile acids | 4 weeks
  plasma microbial metabolites
Concentration of Short chain fatty acids | 4 weeks
  Fecal microbial metabolites
Concentration of urolithins and other ellagitannin-derived metabolites | 4 weeks
  microbial metabolites
Concentration of soluble NADPH oxidase (NOX2) | 4 weeks
  plasma marker oxidative stress
Concentration of uric acid | 4 weeks
  plasma marker oxidative stress
Concentration of total Nitrate/Nitrite and Nitric Oxide related metabolites (RSNO) | 4 weeks
  dietary nitrate and NO metabolites
Concentration of untargeted metabolomics | 4 weeks
  metabolism
Determination of microbial populations | 4 weeks
  stool bacterial population

CONTACTS AND LOCATIONS:
Overall Officials: Carl L Keen, PhD, Principal Investigator — University of California, Davis; Department of Nutrition
Locations (1):
- University of California, Davis; Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/join-this-nutrition-study-of-the-influence-of-honey-flavored-yogurt-on-gut-health-148082/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT04248127/Prot_SAP_000.pdf